CLINICAL TRIAL: NCT00551304
Title: Native Kidney Denervation in Patients With End Stage Renal Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-020 & TP-039
Record Dates: First submitted 2007-10-26; First posted 2007-10-30 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Ardian Catheter

SUMMARY:
To investigate the utility of renal denervation in the treatment of patients with End Stage Renal Disease (ESRD).

ELIGIBILITY:
Inclusion Criteria:

* adult >= 18 years of age
* end stage renal disease, undergoing concurrent dialysis treatment
* poorly controlled blood pressure on at least 2 antihypertensive drugs
* agrees to have the study procedure(s) performed and additional procedures and evaluations, including interventions and follow up visits
* competent and willing to provide written, informed consent to participate in this clinical study.

Exclusion Criteria:

* renal arterial abnormalities
* myocardial infarction, unstable angina pectoris, or a cerebrovascular accident within six (6) months
* hemodynamically significant valvular heart disease
* implantable cardioverter defibrillator (ICD) or pacemaker
* respiratory support.
* pregnant, nursing or planning to be pregnant
* other

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-10

PRIMARY OUTCOMES:
To provide confirmation that renal denervation in ESRD patients is safe and feasible.

SECONDARY OUTCOMES:
To provide evidence of denervation, indication of physiologic response, and assess device performance.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Schlaich, MD, Principal Investigator — The Alfred
Locations (2):
- The Alfred Hospital, Melbourne, Victoria, Australia
- John Paull II Hosptial, Krakow, Poland

REFERENCES:
- [Derived] Schlaich MP, Hering D, Sobotka PA, Krum H, Esler MD. Renal denervation in human hypertension: mechanisms, current findings, and future prospects. Curr Hypertens Rep. 2012 Jun;14(3):247-53. doi: 10.1007/s11906-012-0264-9. PMID 22457244
- [Derived] Hering D, Esler MD, Krum H, Mahfoud F, Bohm M, Sobotka PA, Schlaich MP. Recent advances in the treatment of hypertension. Expert Rev Cardiovasc Ther. 2011 Jun;9(6):729-44. doi: 10.1586/erc.11.71. PMID 21714604
- [Derived] Schlaich MP, Sobotka PA, Krum H, Whitbourn R, Walton A, Esler MD. Renal denervation as a therapeutic approach for hypertension: novel implications for an old concept. Hypertension. 2009 Dec;54(6):1195-201. doi: 10.1161/HYPERTENSIONAHA.109.138610. Epub 2009 Oct 12. No abstract available. PMID 19822798